CLINICAL TRIAL: NCT00380653
Title: A Phase I Pharmacologic Study of Oral Sapacitabine in Patients With Advanced Leukemias or Myelodysplastic Syndromes
Brief Title: Safety and Pharmacology Study of Sapacitabine to Treat Advanced Leukemias or Myelodysplastic Syndromes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cyclacel Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CYC682-05-04
Record Dates: First submitted 2006-09-23; First posted 2006-09-26 (Estimated); Last update posted 2021-12-13 (Actual); Status verified 2021-12

CONDITIONS: Leukemias; Myelodysplastic Syndromes
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes | interventions — sapacitabine

STUDY DESIGN:
Intervention Model Description: The starting dose is (A) 75 mg twice daily x 7 days followed by 14 days of rest or, (B) 375 mg twice daily x 3 consecutive days per week for 2 weeks followed by 7days of rest.
  Evaluated doses in schedule A: 75mg, 100mg, 125mg, 175mg, 225mg, 275mg, 325mg and 375mg Evaluated doses in schedule B: 375mg, 425mg and 475mg

ARMS (2):
- sapacitabine low dose (Experimental): sapacitabine administered every 12 hours for 7 days followed by 14 days of rest or every 12 hours for 3 consecutive days per week for 2 weeks followed by 7 days of rest in patients with advanced leukemias or myelodysplastic syndromes The starting dose is (A) 75 mg twice daily x 7 days followed by 14 days of rest; Evaluated doses: 75mg, 100mg, 125mg, 175mg, 225mg, 275mg, 325mg and 375mg
  Interventions: Drug: sapacitabine
- sapacitabine high dose (Experimental): The starting dose is 375 mg twice daily x 3 consecutive days per week for 2 weeks followed by 7days of rest.
  Evaluated doses: 375mg, 425mg and 475mg
  Interventions: Drug: sapacitabine

INTERVENTIONS:
Drug: sapacitabine
  Other Names: CYC682

SUMMARY:
The goal of this safety/pharmacology study is to determine MTD of sapacitabine when administered in patients with advanced leukemias or myelodysplastic syndromes.

DETAILED DESCRIPTION:
The goal of this study is to find the highest tolerable dose of sapacitabine that can be given to patients with advanced leukemias or myelodysplastic syndromes.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with advanced leukemias or myelodysplastic syndromes defined in section 4.1; Eastern Cooperative Oncology Group performance status 0-2; adequate hepatic and renal function; ability to swallow capsules; be at least 2 weeks from prior chemotherapy, radiation therapy, major surgery or other investigational anticancer therapy; and have recovered from prior toxicities.

Exclusion Criteria:

* Patients with known CNS involvement by leukemia; plan to undergo allogeneic bone marrow transplant within 4 weeks; currently on other investigational agents; uncontrolled intercurrent illnesses; pregnant or lactating women; known to be HIV positive

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2006-01; Primary Completion 2008-11 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose | Through study completion, average of 1 year
  dose limiting toxicities; during first cycle, each cycle is three weeks

CONTACTS AND LOCATIONS:
Overall Officials: Judy H Chiao, MD, Study Director — Cyclacel Pharmaceuticals, Inc.
Locations (1):
- The University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Result] Kantarjian H, Garcia-Manero G, O'Brien S, Faderl S, Ravandi F, Westwood R, Green SR, Chiao JH, Boone PA, Cortes J, Plunkett W. Phase I clinical and pharmacokinetic study of oral sapacitabine in patients with acute leukemia and myelodysplastic syndrome. J Clin Oncol. 2010 Jan 10;28(2):285-91. doi: 10.1200/JCO.2009.25.0209. Epub 2009 Nov 23. PMID 19933907
- See also: Phase I clinical and pharmacokinetic study of oral sapacitabine in patients with acute leukemia and myelodysplastic syndrome. — http://jco.ascopubs.org/content/28/2/285